CLINICAL TRIAL: NCT04312295
Title: The Effects of an ACP Simulation-based Communication Training Program for Nurses Discussing ACP With Chronic Kidney Disease Patients: A Longitudinal Study
Brief Title: ACP Simulation-based Communication Training Program for Nurses Discussing ACP With Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(I)-20150279
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP-SCT program (Experimental): The ACP simulation-based communication training (ACP-SCT)program was designed 12 hours (4hours/week) workshop for nephrology nurses.
  Interventions: Behavioral: ACP-SCT program
- Without ACP-SCT program (No Intervention): The control group only gives the ACP simulation-based communication training program handbook.

INTERVENTIONS:
Behavioral: ACP-SCT program — The ACP-SCT program was designed to improve nurses' knowledge and competence in discussing ACP with Chronic Kidney Disease patients.
  Arms: ACP-SCT program

SUMMARY:
This study was to evaluate the effects of ACP simulation-based communication training program (ACP-SCT program) for nurses to discuss ACP with chronic kidney disease patients

DETAILED DESCRIPTION:
The ACP-SCT program was including three stages, as follows Stage I: To discuss ACP knowledge and law Objective: Opportunity to share experiences, and develop a mutual understanding of the the challenge of ACPdiscussing with CKD patients.

Stage II: communication skills section and Feedback section Objective: 1. To provide a structured approach to managing ACP discussions. 2. Opportunity to practice communication skills in a safe environment 3. Opportunity to discuss their experiences of the training program, and reflect future on their own practice and experience.

ELIGIBILITY:
Inclusion Criteria:

* Participants were nephrology nurses and worked at least one year

Exclusion Criteria:

* Non-nephrology nurses

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
ACP Knowledge Scale | pretest (before training program), Immediate test (after training program), post-test (3 month after training program)
  To evaluate the change of knowledge score for nurses from start of training program to end of training program 3 month later. Nurses' knowledge of discussing ACP will measure using the ACP knowledge Scale developed for this study. This Scale consisting of 20 items; each item consisted of a statement for which a participant could answer ''Yes'' to give 1 point, ''No'' or ''don't know'' to get 0 point. A higher scores indicates more knowledge. Data will analysis using SPSS 22.0 statistical software. Descriptive statistics are calculating as frequencies with percentages and means with standard deviation. Generalized estimating equation (GEE) methods with exchangeable working covariance structure will use to examine group differences in ACP knowledge outcomes, adjusting for changes over time. The GEE provides unbiased estimates of intervention effects.
ACP Confidence Scale | pretest (before training program), Immediate test (after training program), post-test (3 month after training program)
  To evaluate the change of confidence score for nurses from start of training program to end of training program 3 month later. Nurses' self-confidence of communication skills in discussing ACP will measure using the ACP Confidence Scale developed for this study. The instrument consists of 12 items with response options from 0 (not confident at all) to 10(very confident), reflecting an individual's level of confident; higher scores indicates greater confidence. Data will analysis using SPSS 22.0 statistical software. Descriptive statistics are calculating as frequencies with percentages and means with standard deviation. Generalized estimating equation (GEE) methods with exchangeable working covariance structure will use to examine group differences in ACP confidence outcomes, adjusting for changes over time. The GEE provides unbiased estimates of intervention effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jui-O Chen, Mater, Principal Investigator — Tajen University
Locations (1):
- Tajen University, Pingtung City, Yanpu Township, Taiwan

REFERENCES:
- [Derived] Chen JO, Chang SC, Lin CC. The development and pilot testing of an ACP simulation-based communication-training program: Feasibility and acceptability. PLoS One. 2021 Aug 24;16(8):e0254982. doi: 10.1371/journal.pone.0254982. eCollection 2021. PMID 34428209